CLINICAL TRIAL: NCT03838575
Title: A Phase III, Multi-arm, Multi-stage (MAMS), Pragmatic, Blinded (Patient and Outcome Assessor), Multicentre, Randomised Controlled Trial (RCT) With an Internal Pilot, to Evaluate the Use of Several In-theatre Interventions, Used Alone or in Combination, to Reduce SSI Rates in Patients Undergoing Abdominal Surgery.
Brief Title: ROSSINI 2 - Reduction of Surgical Site Infection Using Several Novel Interventions
Acronym: ROSSINI 2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Birmingham (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RG_18-186
Record Dates: First submitted 2019-02-05; First posted 2019-02-12 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-06

CONDITIONS: Surgical Site Infection; Surgical Wound Infection; Surgery--Complications; Surgery
Keywords: SSI; Surgical Site Infection; Infection Prevention; MAMS; Multi-arm, Multi-stage; Pragmatic; Abdominal Surgery; Multicentre; RCT; Pilot; Chlorhexidine; Skin Prep; Iodophor; Drape; Gentamicin; Sponge; Surgery
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: This major, multicentre, multi-arm, multi-stage (MAMS) trial with the opportunity to cease (and introduce) arms would be the first of its kind in a surgical setting. In addition to generating new knowledge in our primary research area, by utilising this advanced design in the context of our relatively simple primary endpoint of SSI, it will also pave the way for future efficient and rapid trials in other aspects of surgical care.
  Please note: In January 2022, following the first interim analysis, arms including intervention 2 - Iodophor-impregnated incise drape (arms C, E, G and H) were closed to recruitment. This means that only 3 interventional arms (4 including the control arm) remain in the trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: ROSSINI 2 is a double blind trial; both the patient and outcome assessor will be blinded to the intraoperative intervention(s). It is not possible to blind the operating surgeon to the intervention allocation.
  The following measures will be taken to ensure concealment of the chosen intervention(s) (blinding):
  * Randomisation in theatre after induction of anaesthesia
  * The intraoperative interventions used will not be documented in the operation notes or in the patient's notes.
  * The skin around the closed wound will be wiped clean using a wet sterile towel at the end of the procedure to prevent unblinding.
  * Clinical follow-up will be conducted by a trained surgeon or a trained member of the local research team who did not participate in the index procedure or surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- A - NONE (Control) (Active Comparator): Any skin preparation of the surgeon's choice may be used in the control arm apart from 2.0% Alcoholic Chlorhexidine Skin Prep.
  No drapes or sponges of any kind may be used.
  Interventions: Other: NONE (Control)
- B - SKIN PREP (Active Comparator): Mechanism: A broad-spectrum antiseptic to clean and prepare the skin prior to surgery.
  Supplier: BD
  Interventions: Drug: 2% alcoholic chlorhexidine skin prep (SKIN PREP)
- C - DRAPE (Other): Please note: In January 2022, following the first interim analysis, arms including intervention 2 - Iodophor-impregnated incise drape (arms C, E, G and H) were closed to recruitment.
  Mechanism: A thin impregnated plastic sheet applied to the prepared skin prior to incision to maintain sterility.
  Supplier: 3M Infection Prevention
  Interventions: Device: Iodophor Antimicrobial Incise Drapes (DRAPE)
- D - SPONGE (Active Comparator): Mechanism: Small absorbable sponges placed into the wound at the time of closure which deliver high concentrations of antibiotic locally to kill pathogens present that may go on to cause SSI.
  Supplier: SERB
  Interventions: Device: Gentamicin-impregnated implants/ sponges (SPONGE)
- E - SKIN PREP and DRAPE (Other): Please note: In January 2022, following the first interim analysis, arms including intervention 2 - Iodophor-impregnated incise drape (arms C, E, G and H) were closed to recruitment.
  See descriptions in single arms (B & C)
  Interventions: Drug: 2% alcoholic chlorhexidine skin prep (SKIN PREP); Device: Iodophor Antimicrobial Incise Drapes (DRAPE)
- F - SKIN PREP and SPONGE (Active Comparator): See descriptions in single arms (B & D)
  Interventions: Drug: 2% alcoholic chlorhexidine skin prep (SKIN PREP); Device: Gentamicin-impregnated implants/ sponges (SPONGE)
- G - DRAPE and SPONGE (Other): Please note: In January 2022, following the first interim analysis, arms including intervention 2 - Iodophor-impregnated incise drape (arms C, E, G and H) were closed to recruitment.
  See descriptions in single arms (C & D)
  Interventions: Device: Iodophor Antimicrobial Incise Drapes (DRAPE); Device: Gentamicin-impregnated implants/ sponges (SPONGE)
- H - SKIN PREP and DRAPE and SPONGE (Other): Please note: In January 2022, following the first interim analysis, arms including intervention 2 - Iodophor-impregnated incise drape (arms C, E, G and H) were closed to recruitment.
  See descriptions in single arms (B, C & D)
  Interventions: Drug: 2% alcoholic chlorhexidine skin prep (SKIN PREP); Device: Iodophor Antimicrobial Incise Drapes (DRAPE); Device: Gentamicin-impregnated implants/ sponges (SPONGE)

INTERVENTIONS:
Drug: 2% alcoholic chlorhexidine skin prep (SKIN PREP) — This intervention describes the preparation of the intact skin incision site immediately prior to incision, using chlorhexidine gluconate (CHG) in an alcohol-based solution, providing durable sterilisation of the surgical field. Pre-prepared applicators will be available for use in this trial (ChloraPrep™ sticks, 2% CHG with 70% isopropyl alcohol, BD Infection Prevention).
  Other Names: Chloraprep
  Arms: B - SKIN PREP; E - SKIN PREP and DRAPE; F - SKIN PREP and SPONGE; H - SKIN PREP and DRAPE and SPONGE
Device: Iodophor Antimicrobial Incise Drapes (DRAPE) — Please note: In January 2022, following the first interim analysis, arms including intervention 2 - Iodophor-impregnated incise drape (arms C, E, G and H) were closed to recruitment.
  This intervention describes the application of a single Iodophor Antimicrobial Incise Drape to be applied topically onto the prepared and draped surgical field by sterile, gloved members of the surgical team before the surgical incision is performed. Only after the skin preparation solution has dried completely can the incise drape be applied.
  Other Names: Ioban Incise Drape
  Arms: C - DRAPE; E - SKIN PREP and DRAPE; G - DRAPE and SPONGE; H - SKIN PREP and DRAPE and SPONGE
Device: Gentamicin-impregnated implants/ sponges (SPONGE) — This intervention describes the implantation of Gentamicin-impregnated collagen implants at the time of fascial closure. Each sponge (10 by 10 cm) contains 280mg of collagen and 130mg of gentamicin. The sponges gradually degrade and the gentamicin solution permeates into surrounding tissues to create a high local antimicrobial concentration within the surgical wound.
  Other Names: Collatamp G
  Arms: D - SPONGE; F - SKIN PREP and SPONGE; G - DRAPE and SPONGE; H - SKIN PREP and DRAPE and SPONGE
Other: NONE (Control) — Any skin preparation of the surgeon's choice may be used in the control arm apart from 2.0% Alcoholic Chlorhexidine Skin Prep.
  No drapes or sponges of any kind may be used.
  Arms: A - NONE (Control)

SUMMARY:
ROSSINI 2 is a phase III, multi-arm, multi-stage (MAMS) pragmatic, blinded (patient and outcome assessor), multicentre, randomised controlled trial (RCT) with an internal pilot, to evaluate the use of several in-theatre interventions, used alone or in combination, to reduce SSI rates in patients undergoing surgery.

DETAILED DESCRIPTION:
The primary objective of ROSSINI 2 is to determine whether several specific in-theatre interventions, used alone or in combination, result in decreased rates of surgical site infection (SSI) up to 30 days post operation in adult patients undergoing abdominal surgery.

At least 60 NHS hospitals in the UK will participate in ROSSINI 2.

Approximately 6610 patients will be required to detect a 5% absolute risk reduction in the intervention arm(s) (15% to 10%; 33% relative reduction) with 85% power.

Initially, the three health technologies that were assessed versus the control arm (standard care) were:

1. 2% alcoholic chlorhexidine skin preparation, versus any other standard skin preparation
2. Iodophor-impregnated incise drape, versus no drape
3. Gentamicin-impregnated implants/ sponge at closure, versus no implant

Please note: In January 2022, following the first interim analysis, arms including intervention 2 - Iodophor-impregnated incise drape (arms C, E, G and H) were closed to recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing colorectal, hepatobiliary, upper GI, urological, vascular, or gynaecological operations
* Patients undergoing abdominal operations (open or laparoscopic extraction site) with a planned incision of at least 5cm.
* Patients aged 16 years or older
* Patients able and willing to undergo a wound assessment at day 30-37 after surgery
* Patients able and willing to give written informed consent
* All contamination strata, including clean, clean-contaminated, contaminated or dirty surgery.
* Patients undergoing planned (elective or expedited) or unplanned (emergency) surgery.

Exclusion Criteria:

* Previous laparotomy within 3 months prior to randomisation
* Known to be pregnant or currently breast feeding
* Operations where the wound is not anticipated to be closed primarily
* Patients with a new or documented allergy/ intolerance to any of the study interventions (chlorhexidine, iodine, collagen or gentamicin) will not be randomised to an arm containing this intervention, but will still be eligible for recruitment to other arms of the study.
* Patients with end-stage renal failure where gentamicin administration would otherwise be contra-indicated (according to local policy) will not be randomised to arms containing the gentamicin-impregnated sponge.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6610 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
SSI rate up to 30 days after surgery as defined according to the 2017 Centers for Disease Control (CDC) and Prevention Criteria. | 30 days post surgery
  The CDC definition will be used in ROSSINI 2 to identify deep incisional or superficial incisional SSIs.

SECONDARY OUTCOMES:
30-day postoperative mortality rate (POMR). | Within 30 days post surgery
  The 30-day postoperative mortality rate (POMR) is determined as death of a patient within the first 30 postoperative days, with day of surgery taken as day 0.
30-day postoperative wound complication rate. | Within 30 days post surgery
  The 30-day postoperative complication rate is determined as the highest level Clavien-Dindo grade complication measured in the first 30 postoperative days, with day of surgery taken as day 0. Any deviation from the normal postoperative course that has an adverse effect on the patient and is not either a treatment failure or sequel, is a complication. The Clavien-Dindo classification determines the severity of a complication based on the therapeutic consequence of that complication.
Serious Adverse Events up to 30 days (wounds or intervention-related only). | Within 30 days post surgery
  The following SAEs (that are related to the use of each intervention (or the control)) should always be recorded and reported (within 24 hours) to the BCTU Trials Office as a SAE, on the
  In-Theatre Form and SAE Form:
  * Death (related to the trial/ intervention(s))
  * Skin reactions
  * Allergic reactions
  * Combustion
  As ROSSINI 2 is a non - CTIMP, BCTU will not be collecting Suspected Unexpected Serious Adverse Reactions (SUSARs). We will however be collecting Related and Unexpected SAEs.
  A Related and Unexpected Serious Adverse Event (RUSAE) means a SAE occurring to a research participant which in the opinion of the Chief Investigator was:
  * 'Related' that is, it resulted from the administration of any of the research procedures, and
  * 'Unexpected' that is, the type of event is not listed in the protocol as an expected occurrence.
Length of hospital stay after surgery as measured from the date of surgery to the date of discharge. | Measured from the date of surgery (Day 0) to the date of discharge (expected to be within 30 days.)
  Length of hospital stay after surgery will be a 'Time to event' outcome, this will be compared between treatment groups using standard survival analysis methods. Kaplan-Meier survival curves will be constructed for visual presentation of time-to-event comparisons. Cox proportional hazard models will be fitted to obtain adjusted treatment effects which will be expressed as hazard ratios with 95% confidence intervals.
Hospital re-admission for wound related complications within 30 days. | Within 30 days post surgery
  Hospital re-admissions for wound related complications within 30 days after surgery will be a 'Time to event' outcome, this will be compared between treatment groups using standard survival analysis methods. Kaplan-Meier survival curves will be constructed for visual presentation of time-to-event comparisons. Cox proportional hazard models will be fitted to obtain adjusted treatment effects which will be expressed as hazard ratios with 95% confidence intervals.
Occurrence of unplanned wound reopening and/or re-operations within 30 days post-operation. | Within 30 days post surgery
  Occurrence of unplanned wound reopening and/or re-operations within 30 days after surgery will be a 'Time to event' outcome, this will be compared between treatment groups using standard survival analysis methods. Kaplan-Meier survival curves will be constructed for visual presentation of time-to-event comparisons. Cox proportional hazard models will be fitted to obtain adjusted treatment effects which will be expressed as hazard ratios with 95% confidence intervals.
Health-related, preference-based quality of life | Baseline, Day 7, Day 30 and if applicable Ongoing SSI (Day 60, 90, 120 etc)
  QoL will be assessed using the widely validated EuroQol EQ-5D-5L questionnaire at baseline (preoperative), as an inpatient (day 7 or at discharge if sooner) and day 30 mirroring the timings of blinded wound assessment.
Cost-effectiveness | To complete at Day 30 and if applicable Ongoing SSI (Day 60, 90, 120 etc)
  Cost effectiveness will be assessed using the Resource Usage Form to collect patient-level health resource usage both in primary and secondary care; reported in QALYs.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Countess of Chester Hospital, Chester

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers.

DOCUMENTS (1):
  • Study Protocol (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT03838575/Prot_000.pdf